CLINICAL TRIAL: NCT05326984
Title: Effect of Metformin on ABCB1 and AMPK Expression in Adolescents With Newly Diagnosed Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General de Mexico (Other Government)
Responsible Party: Principal Investigator, Daniel Ortiz Morales, Head of pediatric hematology & oncology, Hospital General de Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DI/21/505/03/10
Record Dates: First submitted 2022-02-15; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: adolescents; metformin; ABCB1; AMPK
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: The patients are randomized assigned to one of two groups. One group (control group) will receive conventional chemotherapy during remission induction, the other group will receive conventional chemotherapy plus metformin 1000mgm2 per day during the remission induction.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): This subjets will receive conventional chemotherapy alone. The Remission induction chemotherapy includes a steroid pre-phase of 7 days of prednisone 60mgm2SCD. The proper remission induction phase consist in prednisone 60mgm2 daily from day 0 to 28; Vincristine 1.5mgm2 on days 0, 7, 14 and 21; Doxorubicin 25mgm2 on days 0, 7, 21; L-asparaginase 10, 000 Um2 on days 2, 4, 6, 8, 10 and 12. Etoposide 300mgm2 and cytarabine 300mgm2 on days 22, 25 and 29. Intrathecal chemotherapy is administered on days 0, 7, 14 and 21.
- Interventional group (Experimental): This group will receive conventional chemotherapy plus metformin 1000mgm2 per day, with maximum dose of 850mg three times a day, from day -7 to the end of the remission induction period.
  The Remission induction chemotherapy includes a steroid pre-phase of 7 days of prednisone 60mgm2SCD. The proper remission induction phase consist in prednisone 60mgm2 daily from day 0 to 28; Vincristine 1.5mgm2 on days 0, 7, 14 and 21; Doxorubicin 25mgm2 on days 0, 7, 21; L-asparaginase 10, 000 Um2 on days 2, 4, 6, 8, 10 and 12. Etoposide 300mgm2 and cytarabine 300mgm2 on days 22, 25 and 29. Intrathecal chemotherapy is administered on days 0, 7, 14 and 21.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin will be administered orally to the experimental group by randomization at a dose of 1000mgm2 per day, with maximum dose of 850mg three times a day, from day -7 to the end of the remission induction period.
  Arms: Interventional group

SUMMARY:
Acute lymphoblastic leukemia, is the most frequent cancer in children and adolescents. Some genes have been described to produce drug resistance, as ABCB1 probably by lack of activation of AMPK. Some manuscripts have shown that metformin has antitumoral activity, mainly by activation of AMPK.

This is an experimental one center trial, that pretend analyze the effect of metformin at a dose of 1000mgm2 per day, on the expression of the ABCB1 and AMPK genes, when is added to conventional induction remission chemotherapy in newly diagnosed adolescents with acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
Acute lymphoblastic leukemia, is the most frequent cancer in children and adolescents. By now, chemotherapy agent combination achieves remission in more than 90% of patients. But, adolescents have an adverse prognosis compared with children.

The multiple drug resistant genes are well known the cause resistance in different cancers, most important of these genes are the ABCB gene family, specially ABCB1. This resistance is also reported in acute lymphoblastic leukemia. Also changes in AMPK (adenosine triphosphate) gene expression is related to antitumor effects within the cell.

Metformin, a biguanide, has demonstrated that decrease the intracellular ATP levels by AMPK activation, and the blockade of the glycoprotein P, product of the ABCB1 gene. Many reports had described the effect of metformin on different cancer types. In adults, the use of metformin has demonstrated to be useful improving the overall and event free survival, related to low ABCB1/MDR1 (multidrug resistance 1) expression and high AMPK expression.

The investigators propose if the metformin has any effect on ABCB1/MDR1 and AMPK during remission induction phase in adolescents with newly diagnosed Acute Lymphoblastic Leukemia.

Hypothesis: If metformin is added to standard chemotherapy during the remission induction in Mexican adolescents with newly diagnosed acute lymphoblastic leukemia, so the mRNA (messenger ribonucleid acid) expression levels of the ABCB1 gene will decrease and the AMPK gene expression will increase at the end of remission induction.

This study pretends to evaluate the effect of the addition of metformin to a standard chemotherapy regimen in the modification of the expression of the ABCB1 and AMPK genes during the remission induction of newly diagnosed adolescents with acute lymphoblastic leukemia.

Also to describe the expression levels of ABCB1 and AMPK of healthy adolescents and those diagnosed with acute lymphoblastic leukemia. Compare the expression level of those genes at diagnosis and at the end of remission induction; and to compare the global and event free survival based on the initial expression of those genes, and the use of metformin.

The investigators proposed an randomized open clinical trial to compare the modification of the expression of the ABCB1 and AMPK genes in adolescents with newly diagnosed acute lymphoblastic leukemia in patients receiving conventional chemotherapy versus conventional chemotherapy plus metformin 1000 mgm2SC per day during the remission induction phase of the treatment.

All patients with new acute lymphoblastic leukemia between 10 and 21 years old are invited to participate, with informed consent authorized. The exclusion criteria includes patients with previous use of steroids or other chemotherapy, and patients with Down syndrome.

The investigators pretend to enroll 10 patients for each group. After the morphological and cytometry diagnosis confirmation of acute lymphoblastic leukemia, the adolescents are invited to participate with informed consent signed by the patients and legally authorized representative.

The samples are obtain from mononuclear cells from peripheral blood, the total RNA (Ribonuceid acid) are obtain by TRIzol ® (Invitrogen(R) Life Technologies). The integrity and purity of the nucleic acid are determined by spectrophotometry. The RNA is frozen at -80ºC until needed. The DNAc (complementary desoxyribonucelic acid) synthesis is made from 2micrograms of RNA, oligonucleotides, dNTPs, buffer, MgCl2, KCl (potassium chloride), and DTT (dithiothreitol) are added to obtain a final volume of 20micrograms. The mix is incubated at 37ºC for 2 minutes and 1microliter of inverse transcriptase, and incubated for 50 minutes at 37ºC. The qRT-PCR (quantitative Real time-plymerase chain reaction) of the genes is made using the genic expression assay TaqMan®. The expression levels are calculated using the 2-delta-delta-Ct method.

The Remission induction chemotherapy includes a steroid pre-phase of 7 days of prednisone 60 mgm2SCD. The proper remission induction phase consist in prednisone 60 mgm2 daily from day 0 to 28; Vincristine 1.5mgm2 on days 0, 7, 14 and 21; Doxorubicin 25mgm2 on days 0, 7, 21; L-asparaginase 10, 000 Um2 on days 2, 4, 6, 8, 10 and 12. Etoposide 300mgm2 and cytarabine 300mgm2 on days 22, 25 and 29. Intrathecal chemotherapy is administered on days 0, 7, 14 and 21. After the remission induction scheme, bone marrow aspiration is performed to evaluate morphology, if less of 5% of lymphoid blast are reported, the patients continue with consolidation phase with high dose methotrexate and 6 mercaptopurine, and after that the maintenance phase until the end of the protocol.

The intermediate variables are the peripheral blast count on day 0, morphology examination of bone marrow on days 14 and at the end of induction and end of induction MRD (minimal residual disease).

Metformin will be administered to the experimental group by randomization at a dose of 1000mgm2 per day, with maximum dose of 850mg three times a day, from day -7 to the end of the remission induction period. The procurement of the peripheral blood samples for determination of the expression od the genes ABCB1 and AMPK will be made on day -7 and at the end of the remission induction. Follow up of the patient will be done to calculate the global and event free survival.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed adolescents with acute lymphoblastic leukemia by morphology analysis in bine marrow
* Adolescents between 10 and 21 years old
* Participants with the informed consent signed by themselves and the parents or legally authorized representative.

Exclusion Criteria:

* Participants with previous use of any antineoplastic drug
* Down syndrome patients

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-02-09 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Decrease of ABCB1 gene expression | The assessment of ABCB1 gene expression will be made at diagnosis (day -7) and at the end of remission induction phase on day +33
  During the trial ABCB1 gene expression is measure by rt-PCR in mononuclear cells in peripheral blood, at at the beginning of treatment and end of the remission induction
Increase of AMPK gene expression | The assessment of AMPK gene expression will be made at diagnosis (day -7) and at the end of remission induction phase on day +33
  During the trial AMPK gene expression is measure by rt-PCR in mononuclear cells in peripheral blood, at athe beginning and end of the remission induction.

SECONDARY OUTCOMES:
Overall survival | From randomization and initiation of the treatment until the date of death from any cause, assessed up to 2 years
  The probability of being alive after the randomization of the subjects. Is going to be measure by Kaplan Meir method, and compare between the expression of ABCB1 and AMPK genes, and the use of metformin with the log rank statistics.
Event free survival | From randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed upt to 2 years
  The probability of being alive without relapse after randomization of the participants. Will be assess by Kaplan Meir statistics, and compare with log rank.

CONTACTS AND LOCATIONS:
Overall Officials: Adolfo Martinez Tovar, PhD, Study Chair — Hospital General de méxico
Locations (1):
- Hospital General de México, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
The data is going to be coded, and the relation between data and code are only known by the researches and the IRB (institutional review board).

REFERENCES:
- [Background] Smith MA, Seibel NL, Altekruse SF, Ries LA, Melbert DL, O'Leary M, Smith FO, Reaman GH. Outcomes for children and adolescents with cancer: challenges for the twenty-first century. J Clin Oncol. 2010 May 20;28(15):2625-34. doi: 10.1200/JCO.2009.27.0421. Epub 2010 Apr 19. PMID 20404250
- [Background] Rivera-Luna R, Shalkow-Klincovstein J, Velasco-Hidalgo L, Cardenas-Cardos R, Zapata-Tarres M, Olaya-Vargas A, Aguilar-Ortiz MR, Altamirano-Alvarez E, Correa-Gonzalez C, Sanchez-Zubieta F, Pantoja-Guillen F. Descriptive Epidemiology in Mexican children with cancer under an open national public health insurance program. BMC Cancer. 2014 Oct 29;14:790. doi: 10.1186/1471-2407-14-790. PMID 25355045
- [Background] Hunger SP, Lu X, Devidas M, Camitta BM, Gaynon PS, Winick NJ, Reaman GH, Carroll WL. Improved survival for children and adolescents with acute lymphoblastic leukemia between 1990 and 2005: a report from the children's oncology group. J Clin Oncol. 2012 May 10;30(14):1663-9. doi: 10.1200/JCO.2011.37.8018. Epub 2012 Mar 12. PMID 22412151
- [Background] Wolfson JA, Richman JS, Sun CL, Landier W, Leung K, Smith EP, O'Donnell M, Bhatia S. Causes of Inferior Outcome in Adolescents and Young Adults with Acute Lymphoblastic Leukemia: Across Oncology Services and Regardless of Clinical Trial Enrollment. Cancer Epidemiol Biomarkers Prev. 2018 Oct;27(10):1133-1141. doi: 10.1158/1055-9965.EPI-18-0430. Epub 2018 Sep 27. PMID 30262597
- [Background] Dean M, Rzhetsky A, Allikmets R. The human ATP-binding cassette (ABC) transporter superfamily. Genome Res. 2001 Jul;11(7):1156-66. doi: 10.1101/gr.184901. PMID 11435397
- [Background] Szakacs G, Paterson JK, Ludwig JA, Booth-Genthe C, Gottesman MM. Targeting multidrug resistance in cancer. Nat Rev Drug Discov. 2006 Mar;5(3):219-34. doi: 10.1038/nrd1984. PMID 16518375
- [Background] Rahgozar S, Moafi A, Abedi M, Entezar-E-Ghaem M, Moshtaghian J, Ghaedi K, Esmaeili A, Montazeri F. mRNA expression profile of multidrug-resistant genes in acute lymphoblastic leukemia of children, a prognostic value for ABCA3 and ABCA2. Cancer Biol Ther. 2014 Jan;15(1):35-41. doi: 10.4161/cbt.26603. Epub 2013 Oct 21. PMID 24145140
- [Background] Giovannucci E, Harlan DM, Archer MC, Bergenstal RM, Gapstur SM, Habel LA, Pollak M, Regensteiner JG, Yee D. Diabetes and cancer: a consensus report. Diabetes Care. 2010 Jul;33(7):1674-85. doi: 10.2337/dc10-0666. PMID 20587728
- [Background] Trucco M, Barredo JC, Goldberg J, Leclerc GM, Hale GA, Gill J, Setty B, Smith T, Lush R, Lee JK, Reed DR. A phase I window, dose escalating and safety trial of metformin in combination with induction chemotherapy in relapsed refractory acute lymphoblastic leukemia: Metformin with induction chemotherapy of vincristine, dexamethasone, PEG-asparaginase, and doxorubicin. Pediatr Blood Cancer. 2018 Sep;65(9):e27224. doi: 10.1002/pbc.27224. Epub 2018 Jun 1. PMID 29856514
- [Background] Leclerc GM, Leclerc GJ, Kuznetsov JN, DeSalvo J, Barredo JC. Metformin induces apoptosis through AMPK-dependent inhibition of UPR signaling in ALL lymphoblasts. PLoS One. 2013 Aug 23;8(8):e74420. doi: 10.1371/journal.pone.0074420. eCollection 2013. PMID 24009772
- [Background] Dowling RJ, Niraula S, Stambolic V, Goodwin PJ. Metformin in cancer: translational challenges. J Mol Endocrinol. 2012 Mar 29;48(3):R31-43. doi: 10.1530/JME-12-0007. Print 2012 Jun. PMID 22355097
- [Background] Kim HG, Hien TT, Han EH, Hwang YP, Choi JH, Kang KW, Kwon KI, Kim BH, Kim SK, Song GY, Jeong TC, Jeong HG. Metformin inhibits P-glycoprotein expression via the NF-kappaB pathway and CRE transcriptional activity through AMPK activation. Br J Pharmacol. 2011 Mar;162(5):1096-108. doi: 10.1111/j.1476-5381.2010.01101.x. PMID 21054339

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/84/NCT05326984/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/84/NCT05326984/ICF_001.pdf